CLINICAL TRIAL: NCT02802527
Title: Percutaneous Tracheostomy - Systematic Comparison Among Two Methods: Bronchoscopy Guided Tracheostomy, and Direct Laryngoscopy Tracheostomy
Brief Title: Percutaneous Tracheostomy - Systematic Comparison Among Two Methods
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TRACH- HMO-CTIL
Record Dates: First submitted 2016-04-13; First posted 2016-06-16 (Estimated); Last update posted 2016-06-16 (Estimated); Status verified 2016-04

CONDITIONS: Other Tracheostomy Complication

ARMS (2):
- Bronchoscopy Guided (Other): Percutaneous tracheostomy will be guided by bronchoscopy. Initially, the tube will be placed according to the desired height observed by the bronchoscope, phase two will be tracheal perforation by a needle under trans illumination and real-time view on the income of the needle and the passage of the guide wire.
  Interventions: Procedure: Percutaneous Tracheostomy
- Direct Laryngoscopy (Other): Performing percutaneous tracheostomy by placing the tube higher up, near the vocal cords by direct laryngoscopy. In the second stage tracheal perforation by a needle will be carried out by palpation of the anatomical placement of the neck.
  Interventions: Procedure: Percutaneous Tracheostomy

INTERVENTIONS:
Procedure: Percutaneous Tracheostomy

SUMMARY:
Percutaneous tracheostomy is routinely performed in most intensive care units in the world.Several studies have shown that the procedure is safe and economically efficient in comparison to open surgical operation in the operating room.

In the investigator's institution as in a number of institutions in the country and abroad, it is acceptable to perform the operation either by withdrawing the endotracheal tube to a position near the vocal cords by direct laryngoscopy and then puncturing the trachea with a needle distal to the endotracheal tube, prior to carrying out the PDT, by location of the anatomy by palpation of the neck, or alternatively by doing the entire procedure under bronchoscopic guidance.

So far, no systematic comparison has been made between the two methods ie PDT without bronchoscopy versus PDT with bronchoscopy.

DETAILED DESCRIPTION:
Introduction Percutaneous dilatational tracheostomy (PDT) is routinely performed in most intensive care units in the world for a number of indications, such as: airway obstruction, need for long-term respiratory support, improvement in trachea-bronchial toilet, prophylaxis before head and neck procedures, cases of severe obstructive sleep apnea and poor neurological state.

Several studies have shown that the procedure is safe and economically efficient in comparison to open surgical tracheostomy in the operating room.

In many places around the world it is customary to perform the procedure under direct visions via a bronchoscope to prevent damage to adjacent structures, ensure correct position of the tracheostomy tube, avoid damage to the posterior wall of the trachea and to confirm the final position of the tube. However, the use of a bronchoscope depends on the availability of the equipment and knowledge and skill of the operator. Use of the bronchoscope during the procedure may also result in complications such as temporary occlusion of the trachea and hypercarbia and increased duration of the procedure. Maintenance of the bronchoscope also carries associated costs (disinfection, replacement, etc.).

A retrospective review of 243 percutaneous tracheostomies done in trauma patients between January 2007 and December 2010 in whom 78 (32%) was performed with a bronchoscope and 168 (68%) without, found no differences between the groups 4.

Another retrospective study 5 looking only at percutaneous tracheostomies done without bronchoscopic guidance, analyzed 300 PDTs showed that 26 patients (8.6%) had complications, including: 2 (0.6%) patients deteriorated neurologically and 2 (0.6%) deaths were observed within 24 h following procedure. The median operating time was 3.5 min (range, 2.5-8 min). There were no cannula placement problems in any case . A retrospective study looking at 512 bronchoscopy guided procedures over 10 years concluded that: Eighteen patients (3.5%) presented procedural complications. Five patients experienced transient desaturation, 4 presented low blood pressure related to sedation, and 9 presented minor bleeding, but none required a transfusion. No serious complications or deaths associated with the procedure were recorded. Eleven patients (2.1%) presented post-operative complications. Seven presented minor and transitory bleeding of the percutaneous tracheostomy stoma, 2 suffered displacement of the tracheostomy cannula, and 2 developed a superficial infection of the stoma.

In the investigator's institution as in a number of institutions in the country and abroad, it is acceptable to perform the operation either by withdrawing the endotracheal tube to a position near the vocal cords by direct laryngoscopy and then puncturing the trachea with a needle distal to the endotracheal tube, prior to carrying out the PDT, by location of the anatomy by palpation of the neck, or alternatively by doing the entire procedure under bronchoscopic guidance.

So far, no systematic comparison has been made between the two methods ie PDT without bronchoscopy versus PDT with bronchoscopy.

ELIGIBILITY:
Inclusion Criteria:

* All intubated patients with various injuries requiring percutaneous tracheostomy (in- house and out- house patients)
* Minimal age 18

Exclusion Criteria:

* No patient consent for participation
* Anatomical problem which does not allow for percutaneous tracheostomy and requires open procedure in the operating room

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2016-07; Primary Completion 2019-05 (Estimated)

PRIMARY OUTCOMES:
A systematic comparison among the two methods of percutaneous tracheostomy in terms of safety: minor and major periprocedural morbidity. | 30 days

SECONDARY OUTCOMES:
Periprocedural Mortality. | 30 days.
Post procedural ICU & Hospital length of stay. | 30 days.
Complication rate comparison of PDT done in the ICU to PDT done in locations other than the ICU. | 30 days.
Procedure's length. | 60 minutes